CLINICAL TRIAL: NCT04981860
Title: Comparison of Conjunctival Antimicrobial Activity and Patient Comfort Between Topical Hypochlorous Acid (Avenova) and Betadine
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: sample microbiologic results where not consistent
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Jorge Fortun, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200815
Record Dates: First submitted 2021-07-27; First posted 2021-07-29 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Eye Infections, Bacterial
MeSH Terms: conditions — Eye Infections, Bacterial | interventions — Povidone-Iodine; Hypochlorous Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Treatment naïve participants First Group L (Experimental): Treatment naïve participants randomized to receive Betadine on the left eye and Avenova on the right Eye
  Interventions: Drug: Betadine; Drug: Avenova
- Treatment naïve participants Second Group R (Experimental): Treatment naïve participants randomized to receive Avenova on the left eye and Betadine on the right Eye
  Interventions: Drug: Betadine; Drug: Avenova
- Participants undergoing intravitreal injection First Group L (Experimental): Participants undergoing intravitreal injection will receive betadine in the eye that is receiving injections and Avenova in the other eye. Group L are patients that are having intravitreal injections and will receive betadine in the left eye and Avenova in the right eye.
  Interventions: Drug: Betadine; Drug: Avenova
- Participants undergoing intravitreal injection Second Group R (Experimental): Participants undergoing intravitreal injection will receive betadine in the eye that is receiving injections and Avenova in the other eye. Group R are patients that are having intravitreal injections and will receive betadine in the right eye and Avenova in the left eye.
  Interventions: Drug: Betadine; Drug: Avenova

INTERVENTIONS:
Drug: Betadine — One drop of 5% Betadine will be administered to the inferior conjunctiva of the eye
  Other Names: Povidone Iodine
Drug: Avenova — One drop of 0.01% Avenova will be administered to the inferior conjunctiva of the left eye
  Other Names: Hypochlorous Acid

SUMMARY:
The purpose of this research study is to find out how Avenova (0.01 % hypochlorous acid) works compared to Betadine (Povidone iodide) for reducing bacteria and patient discomfort in the eyes.

DETAILED DESCRIPTION:
About two percent of the population have an iodine allergy 1. A percentage of this population will also have a reaction to iodine-containing agents, including povidone iodine (PI) (Betadine®), which is the current standard of care for anti-septic preparation for conjunctival procedures. Despite being known to have a toxic effect on the cornea 2 and causing allergic reactions in some individuals, povidone Iodine (PI) (Betadine®) is still the most commonly used antiseptic agent for surgical scrub. Currently, there are no equivalent alternative prep agents available, although chlorhexidine has occasionally served as an alternative to povidone iodine (PI) (Betadine®) with variable results 2. Some studies have reported significantly less pain in patients prepped with chlorhexidine compared to povidone iodine (PI) (Betadine®) 2, and other studies have demonstrated that chlorhexidine has equal efficacy to povidone iodine (PI)(Betadine®) in decreasing the colony forming units of microbes both in vitro and in vivo 3. Although there have been no known reported allergies to chlorhexidine, it is known to be toxic to the cornea (leading to severe keratitis) and has proven to be less effective against methicillin-resistant Staphylococcus aureus(MRSA) 4.

The use of 0.01% hypochlorous acid (HOCl) in saline solution as an antiseptic agent has been gaining popularity as a possible alternative to povidone iodine (PI) (Betadine®). Hypochlorous acid (HOCl) is produced in vivo by neutrophils and causes oxidation of microbial nucleotides and inactivation of microbial enzymes, leading to cell death. Hypochlorous acid (HOCl) has a faster optimal kill-time for flora common to the eye 4, and has proven to be non-cytotoxic and well tolerated for continuous use 4,5,6. In vitro studies of 0.01% hypochlorous acid (HOCl) were found to have equal or more efficacious antiseptic properties compared with povidone iodine (PI) (Betadine®) and other potential antiseptic agents including chlorohexidine and isopropyl alcohol 4.

Currently, two concentrations of HOCl are available for commercial use: AvenovaTM with Neutrox™ (0.01% HOCl) and an over the counter product (0.02% HOCl). Both concentrations are used to treat blepharitis. Debabov et al5 presented toxicity data concluding that 0.01% hypochlorous acid (HOCl) (Avenova™ with Neutrox™) proved to be non-cytotoxic in comparison to the 0.02% hypochlorous acid (HOCl) product which was cytotoxic thus supporting the potential benefit of HOCl.

Stroman et al6 2017 concludes that hypochlorous acid (HOCl)in saline solution reduced bacterial colony load significantly without altering the variation of remaining bacterial species. Additionally, hypochlorous acid (HOCl) has been shown to reduce the population of bacterial and fungal species common to the lids and lashes by ≥ 99.9% 7. Despite the use of hypochlorous acid (HOCl) as a topical antiseptic on the eyelid, there have been no reports of its use as an antiseptic agent for conjunctival procedures. Many studies have confirmed that flora of the eyelid and eyelash only differ in their concentrations 8. Since hypochlorous acid (HOCl) has been found to be effective in reducing colony forming units and since the flora species of the conjunctiva, eyelid and eyelashes are equivalent, we propose that hypochlorous acid (HOCl) may serve as an alternative to povidone iodine (PI) (Betadine®) as a conjunctival procedure prep agent. Considering there were no reported negative side effects of hypochlorous acid (HOCl) contact with the eye, hypochlorous acid (HOCl) may prove to be a non-inferior alternative to povidone iodine (PI) (Betadine®). This may result in lower irritation and toxicity compared to povidone iodine (PI) (Betadine®)

ELIGIBILITY:
Inclusion criteria:

Treatment Naïve patients:

- Any patient who is able to give consent for the study and did not receive an intravitreal injection in the past 6 months

Patients receiving injections:

- Patient currently undergoing treatment for which he/she receives a intravitreal injection in one eye.

Exclusion Criteria:

Treatment Naïve patients:

* Intravitreal injections in the past 6 months
* Use of eye drops for treatment of glaucoma in the past 6 months
* Use of eye drops with antibiotics or steroids in the past 6 months

Patients receiving injections:

* Patient receiving injections in both eyes
* Use of eye drops for treatment of glaucoma in the past 6 months
* Use of eye drops with antibiotics or steroids in the past 6 months
* Have any condition that, in the opinion of the investigator, would compromise the well-being of the patient or the study or prevent the patient from meeting or performing study requirements.

For both groups:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of bacterial Colony Forming Units (CFU) | Day 1
  As assessed from sterile culture swab applied to the eye

SECONDARY OUTCOMES:
Change in Post Exposure Symptom Severity Scale | Baseline, Day 2
  The Post exposure questionnaire has a total score ranging from 1 to 10 with a higher score indicating greater pain

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Fortun, MD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - Bascom Palmer Eye Institute, Palm Beach Gardens, Florida
  - Medical Center Ophthalmology Associates, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No